CLINICAL TRIAL: NCT04294147
Title: A Phase 4 Single-Blind Study of Gastrointestinal Transit Time in Adult Patients With Migraine Before and After Initiation of a mAb CGRP Antagonist
Brief Title: A Study of Gastrointestinal Emptying Time in Adult Participants With Migraine Before and After Start of a mAb CGRP Antagonist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17590; I5Q-MC-CGBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-03-02; First posted 2020-03-03 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Migraine
Keywords: prevention; prophylaxis; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — galcanezumab; erenumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Galcanezumab (Experimental): Participants received a single subcutaneous (SC) dose of 240 milligram (mg) Galcanezumab.
  Interventions: Drug: Galcanezumab
- Erenumab (Active Comparator): Participants received a single SC dose of 140 mg Erenumab.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
  Arms: Galcanezumab
Drug: Erenumab — Administered SC
  Arms: Erenumab

SUMMARY:
The purpose of this study is to measure the gastrointestinal emptying time using the wireless motility capsule (WMC) technology (FDA approved SmartPill™) in adult participants with migraine who are taking a monoclonal antibody (mAb) calcitonin gene-related peptide (CGRP) antagonist called galcanezumab or erenumab.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine, with or without aura, as determined by the study investigator and in consideration of International Headache Society International Classification of Headache Disorders - 3rd edition guidelines (ICHD-3 2018)
* Have a frequency of less than 15 monthly headache days of which up to 14 can be migraine headache days.
* Participants can be on no more than 1 other migraine preventive treatment (except for tricyclic antidepressants and verapamil which are not allowed) as long as: that participant has had a stable dose of the oral migraine preventive treatment for a minimum of 2 months or participants have received onabotulinumtoxinA for a minimum of 2 cycles prior to screening

Exclusion Criteria:

* Participants with a history of gastric bezoars, swallowing disorders, severe dysphagia to food or pills, suspected or known strictures, fistulas, or physiological/mechanical GI obstruction
* History of any abdominal surgery within the past 3 months or GI surgery with the exception of cholecystectomy, appendectomy, or Nissen fundoplication
* History of irritable bowel syndrome (IBS), chronic constipation, Crohn's disease, celiac disease, ulcerative colitis, or diverticulitis
* Participants with type 1 or type 2 diabetes
* Participants with cardiac pacemakers or other implanted or portable electromechanical device
* Participants with a body mass index of ≥40 kilograms per square meter (kg/m²)
* Women who are pregnant or nursing
* Participants currently on mAb CGRP antagonists or have received a mAb CGRP antagonist within the past 6 months prior to visit 1
* Participants who have received an oral CGRP antagonist (gepant) in the last 14 days prior to Visit 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Clinical Research Institute LLC, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - CMR of Greater New Haven, Waterbury, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Gastrointestinal Emptying Time in Adult Participants With Migraine Before and After Start of a CGRP Antagonist — https://trials.lillytrialguide.com/en-US/trial/1yGB1p2tvaIcLCeMb8TZmI

RESULTS

PARTICIPANT FLOW:
Groups:
- 140 mg Erenumab SC: Participants received a single subcutaneous (SC) dose of 140 milligram (mg) Erenumab.
- 240 mg Galcanezumab SC: Participants received a single SC dose of 240 mg Galcanezumab.
Period: Overall Study
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Started | 32 | 33
Received at Least One Dose of Study Drug | 32 | 33
Completed | 30 | 33
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 140 mg Erenumab SC: Participants received a single SC dose of 140 mg Erenumab.
- Total: Total of all reporting groups
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.4) | 38 (9.5) | 39.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 27
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 6 | 10
  White | 23 | 26 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 33 | 65
Colonic transit time [Mean (Standard Deviation); unit: hours] | 31.5 (28.1) | 28.3 (24.1) | 29.9 (26.0)
Whole Gut Transit Time [Mean (Standard Deviation); unit: hours] | 41.9 (30.3) | 42.3 (29.8) | 42.1 (29.8)
Gastric Emptying Time [Mean (Standard Deviation); unit: hours] | 5.3 (6.3) | 9.3 (17.4) | 7.3 (13.2)
Small Intestine Bowel Transit Time [Mean (Standard Deviation); unit: hours] | 5.1 (1.6) | 4.7 (2.2) | 4.9 (1.9)
Combined Small and Large Intestine Bowel Transit Time [Mean (Standard Deviation); unit: hours] | 36.6 (28.6) | 33.0 (24.7) | 34.8 (26.6)
Motility Index (MI) by Quartile in the Colon [Mean (Standard Deviation); unit: motility index] — Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline MI assessments for each quartile in the colon.
  motility index
    Quartile 1 of Colon: number analyzed (Participants) | 28 | 31 | 59
    Quartile 1 of Colon | 12.352 (2.8544) | 12.201 (2.7862) | 12.2765 (2.8203)
    Quartile 2 of Colon: number analyzed (Participants) | 28 | 31 | 59
    Quartile 2 of Colon | 12.869 (3.0315) | 12.444 (3.0525) | 12.6565 (3.042)
    Quartile 3 of Colon: number analyzed (Participants) | 28 | 31 | 59
    Quartile 3 of Colon | 12.408 (4.0960) | 12.318 (3.9021) | 12.363 (3.99905)
    Quartile 4 of Colon: number analyzed (Participants) | 28 | 31 | 59
    Quartile 4 of Colon | 14.381 (2.1097) | 13.245 (2.2947) | 13.813 (2.2022)
Gastrointestinal Symptom Rating Scale [Mean (Standard Deviation); unit: score on a scale]
  Abdominal pain syndrome | 1.2 (0.5) | 1.2 (0.3) | 1.2 (0.4)
  Reflux syndrome | 1.1 (0.3) | 1.1 (0.3) | 1.1 (0.3)
  Indigestion syndrome | 1.2 (0.3) | 1.3 (0.5) | 1.2 (0.4)
  Constipation syndrome | 1.1 (0.1) | 1.1 (0.2) | 1.1 (0.2)
  Diarrhea syndrome | 1.1 (0.3) | 1.2 (0.4) | 1.2 (0.4)
Bristol Stool Form Scale [Mean (Standard Deviation); unit: score on a scale] | 3.6 (0.9) | 3.8 (1.1) | 3.7 (1.0)
Weekly spontaneous bowel movements (SBMs) [Mean (Standard Deviation); unit: SBMs per week] | 8.6 (3.7) | 9.2 (5.7) | 8.9 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Colonic Transit Time (CTT) at Week 2
Description: Least squares (LS) mean change from baseline was calculated using analysis of covariance (ANCOVA) model with categorical effects of treatment, pooled investigative site, Body mass index (BMI) category (<30kg/m2, ≥30 kg/m2) and baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days) as well as the continuous baseline CTT (hours). A negative change from baseline indicates a decrease in CTT and a positive change from baseline indicate an increase in CTT.
Time Frame: Baseline, Week 2
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline CTT assessments.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 28 | 31
hours | 5.752 (5.7234) | -5.348 (5.4177)

2. Secondary Outcome: Change From Baseline in Whole Gut Transit Time (WGTT) at Week 2
Description: Least squares (LS) mean change from baseline was calculated using ANCOVA model with categorical effects of treatment, pooled investigative site, Body mass index (BMI) category (<30kg/m2, ≥30 kg/m2) and baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days) as well as the continuous baseline WGTT (hours). A negative change from baseline indicates a decrease in WGTT and a positive change from baseline indicate an increase in WGTT.
Time Frame: Baseline, Week 2
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline WGTT assessments.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 28 | 31
hours | 4.123 (5.9808) | -7.043 (5.6307)

3. Secondary Outcome: Change From Baseline in Gastric Emptying Time (GET) at Week 2
Description: Least squares (LS) mean change from baseline was calculated using ANCOVA model with categorical effects of treatment, pooled investigative site, Body mass index (BMI) category (<30kg/m2, ≥30 kg/m2) and baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days) as well as the continuous baseline GET (hours). A negative change from baseline indicates a decrease in GET and a positive change from baseline indicate an increase in GET.
Time Frame: Baseline, Week 2
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline GET assessments.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 28 | 31
hours | -1.320 (1.0299) | -0.582 (0.9691)

4. Secondary Outcome: Change From Baseline in Small Intestine Bowel Transit Time (SBTT) at Week 2
Description: Least squares (LS) mean change from baseline was calculated using ANCOVA model with categorical effects of treatment, pooled investigative site, Body mass index (BMI) category (<30kg/m2, ≥30 kg/m2) and baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days) as well as the continuous baseline SBTT (hours). A negative change from baseline indicates a decrease in SBTT and a positive change from baseline indicate an increase in SBTT.
Time Frame: Baseline, Week 2
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline SBTT assessments.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 28 | 31
hours | -0.551 (0.3138) | -0.719 (0.2935)

5. Secondary Outcome: Change From Baseline in Combined Small and Large Intestine Bowel Transit Time (SLBTT) at Week 2
Description: Least squares (LS) mean change from baseline was calculated using ANCOVA model with categorical effects of treatment, pooled investigative site, Body mass index (BMI) category (<30kg/m2, ≥30 kg/m2) and baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days) as well as the continuous baseline SLBTT (hours). A negative change from baseline indicates a decrease in SLBTT and a positive change from baseline indicate an increase in SLBTT.
Time Frame: Baseline, Week 2
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline SLBTT assessments.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 28 | 31
hours | 5.150 (5.6590) | -5.957 (5.3549)

6. Secondary Outcome: Change From Baseline in Motility Index by Quartile in the Colon at Week 2
Description: Motility index (MI) is a calculated outcome, based on the formula: In (Number of contractions x Σpressure amplitudes +1) where ln = natural logorithm, Σ = Sum. Least squares (LS) mean change from baseline was calculated using ANCOVA model with categorical effects of treatment, pooled investigative site, Body mass index (BMI) category (<30kg/m2, ≥30 kg/m2) and baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days) as well as the continuous baseline MI. A negative change from baseline indicates a decrease in colonic contractions or pressure or both, and a positive change from baseline indicates an increase in colonic contractions or pressure or both.
Time Frame: Baseline, Week 2
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline MI assessments for each quartile in the colon.
Measure: Least Squares Mean (Standard Error); unit: motility index
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 28 | 31
motility index
  Quartile 1 of Colon | 1.111 (0.5226) | 0.367 (0.4912)
  Quartile 2 of Colon | 0.218 (0.7258) | -0.251 (0.6813)
  Quartile 3 of Colon | 0.926 (0.7477) | -0.298 (0.7016)
  Quartile 4 of Colon | 0.489 (0.4723) | -0.035 (0.4445)

7. Secondary Outcome: Change From Baseline in Gastrointestinal (GI) Symptom Rating Scale (GSRS) at Weeks 2 and 4
Description: GSRS is a validated 15-item questionnaire that evaluates the common symptoms of GI disorders. It has five subscales: abdominal pain (abdominal pain, hunger pains, nausea), reflux (heartburn, acid reflux), indigestion (rumbling, bloating, belching, and increased flatus/breaking wind), constipation (constipation, hard stools, and sensation of not completely emptying the bowels), and diarrhea (diarrhea, loose stools, urgent need to have a bowel movement) syndromes. Subscale scores range from 1 to 7. Higher scores indicate greater severity of symptoms. LS mean change from baseline was calculated using mixed effects model for repeated measures (MMRM) with fixed categorical effects of treatment, pooled investigative site, BMI category (<30kg/m2, ≥30 kg/m2), baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days), week, and treatment-by-week interaction, as well as the continuous fixed covariates of baseline value and baseline-by-week interaction.
Time Frame: Baseline, Week 2, Week 4
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline GSRS assessments.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 32 | 33
score on a scale
  Abdominal pain syndrome - Week 2 | -0.041 (0.0826) | 0.022 (0.0799)
  Abdominal pain syndrome - Week 4: number analyzed (Participants) | 30 | 33
  Abdominal pain syndrome - Week 4 | -0.090 (0.0748) | 0.071 (0.0713)
  Reflux syndrome - Week 2 | -0.042 (0.0756) | 0.074 (0.0729)
  Reflux syndrome - Week 4: number analyzed (Participants) | 30 | 33
  Reflux syndrome - Week 4 | 0.078 (0.0862) | 0.17 (0.082)
  Indigestion syndrome - Week 2 | 0.026 (0.0844) | -0.011 (0.0814)
  Indigestion syndrome - Week 4: number analyzed (Participants) | 30 | 33
  Indigestion syndrome - Week 4 | 0.005 (0.0955) | 0.20 (0.091)
  constipation syndrome - Week 2 | 0.41 (0.153) | 0.38 (0.148)
  constipation syndrome - Week 4: number analyzed (Participants) | 30 | 33
  constipation syndrome - Week 4 | 0.25 (0.161) | 0.43 (0.153)
  Diarrhea syndrome - Week 2 | -0.076 (0.0367) | -0.063 (0.0352)
  Diarrhea syndrome - Week 4: number analyzed (Participants) | 30 | 33
  Diarrhea syndrome - Week 4 | -0.057 (0.0852) | 0.072 (0.0807)

8. Secondary Outcome: Change From Baseline in Bristol Stool Form Scale (BSFS) at Weeks 2 and 4
Description: The BSFS is a 7-point ordinal scale which classifies the type of bowel movement based on the appearance of stool. Score 1, 2 indicate constipation (harder stools); 6, 7 indicate diarrhea (loose/liquid stools ); 3 to 5 are considered normal. A better score would trend toward the middle of the scale (3 to 5), while scores at either end of the scale correspond to worse outcomes. LS mean change from baseline was calculated using mixed effects model for repeated measures (MMRM) with fixed categorical effects of treatment, pooled investigative site, BMI category (<30kg/m2, ≥30 kg/m2), baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days), week, and treatment-by-week interaction, as well as the continuous fixed covariates of baseline value and baseline-by-week interaction.
Time Frame: Baseline, Week 2, Week 4
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline BSFS assessments.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 32 | 33
score on a scale
  Week 2 | -0.44 (0.163) | -0.040 (0.1554)
  Week 4: number analyzed (Participants) | 30 | 33
  Week 4 | -0.48 (0.182) | 0.023 (0.1710)

9. Secondary Outcome: Change From Baseline in the Weekly Spontaneous Bowel Movements (SBMs) at Weeks 2 and 4
Description: Weekly SBM is the number of spontaneous (un-aided by laxatives, enemas, or suppositories) bowel movements that a participant has had in the past 7 days. LS mean change from baseline was calculated using mixed effects model for repeated measures (MMRM) with fixed categorical effects of treatment, pooled investigative site, BMI category (<30kg/m2, ≥30 kg/m2), baseline migraine frequency (<8 migraine headache days, ≥8 migraine headache days), week, and treatment-by-week interaction, as well as the continuous fixed covariates of baseline value and baseline-by-week interaction. A negative change from baseline indicates a decrease in weekly SBMs, and a positive change from baseline indicates an increase in weekly SBMs.
Time Frame: Baseline, Week 2, Week 4
Population: All randomized participants who received at least one dose of study drug and had baseline, post-baseline weekly SBM assessments.
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 32 | 33
SBMs per week
  Week 2 | -1.28 (0.537) | 0.31 (0.517)
  Week 4: number analyzed (Participants) | 30 | 33
  Week 4 | -1.13 (0.511) | 0.54 (0.484)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To 28 Days)
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 140 mg Erenumab SC | 240 mg Galcanezumab SC
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 7/32 | 3/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 140 mg Erenumab SC (N=32) | 240 mg Galcanezumab SC (N=33)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04294147/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT04294147/SAP_001.pdf